CLINICAL TRIAL: NCT04159779
Title: Clinical Outcomes of Chronic Lymphocytic Leukemia (CLL) Patients Treated With Venetoclax in Routine Clinical Settings in Greece
Brief Title: A Study of Clinical Outcomes in Chronic Lymphocytic Leukemia (CLL) Patients Treated With Venetoclax in Greece
Status: Active, not recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P19-568
Record Dates: First submitted 2019-11-08; First posted 2019-11-12 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia Venetoclax Relapsed/Refractory
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Venetoclax Participants: Participants for whom the treating physician has decided to treat with venetoclax before enrollment in this study.

SUMMARY:
This study is being done to evaluate the clinical outcomes of Chronic Lymphocytic Leukemia (CLL) participants treated with venetoclax as routine standard of care in Greece. The decision to treat with venetoclax is made by the participant's physician prior to being offered enrollment in this study.

The objectives of this study include determining overall response rate, assessing safety information, analyzing patient profiles and disease characteristics and participant quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Chronic Lymphocytic Leukemia (CLL) according to the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria
* Eligible to receive venetoclax as per local label
* Physician has decided to initiate CLL treatment with venetoclax and the decision to treat is made by the physician in accordance with the local label prior to any decision to approach the participant about the study
* Participant has been fully informed verbally and in writing about the study and does not object to their data being processed or subjected to data quality control

Exclusion Criteria:

* Prescribed or treated with venetoclax outside of marketing authorization
* Currently participating in, or previously participated within 30 days prior to venetoclax start, in any other interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll adult participants (age >=18) with confirmed diagnosis of Relapse/Refractory Chronic Lymphocytic Leukemia being treated with venetoclax in Greece as part of routine standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2020-01-13 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | At Month 12
  Defined by the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) Guidelines and includes partial response (PR), nodular partial response (nPR), complete response with incomplete bone marrow recovery (CRi), and complete response (CR).

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to Month 36
  Defined by the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) Guidelines.
Complete Response (CR) | Up to Month 36
  Defined by the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) Guidelines.
Complete Response with Incomplete Bone Marrow Recovery (CRi) Rate | Up to Month 36
  Defined by the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) Guidelines.
Nodule Partial Response (nPR) Rate | Up to Month 36
  Defined by the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) Guidelines.
Partial Response (PR) Rate | Up to Month 36
  Defined by the International Workshop on Chronic Lymphocytic Leukemia (iwCLL).
Percentage of Participants With Disease Progression or Death | Up to Month 36
  Disease progression as Assessed by the Investigator using International Workshop on Chronic Lymphocytic Leukemia (iwCLL) Guidelines.
Progression Free Survival (PFS) | Up to Month 36
  Defined as the time between the date of first venetoclax intake and the date of the first assessment documenting progression or death (from any cause).
Overall Survival (OS) | Up to Month 36
  Defined as the time from first venetoclax intake to death from any cause.
Treatment Duration | Up to Month 36
  Overall treatment duration of venetoclax.
Time to Progression (TTP) | Up to Month 36
  Defined as the period from first venetoclax intake until objective disease progression (until disease progression or death due to progression, whichever occurs first).
Change in Patient Reported Outcomes | From Baseline (Week 0) Up to Month 36
  The 5-Level EuroQol Group Questionnaire (EQ-5D-5L) is a standardized instrument used to measure health-related quality of life that can be used in a wide range of health conditions and treatments.
Percentage of Participants with Undetectable Minimal Residual Disease (uMRD) | Up to Month 36
  Determined by assessment of peripheral blood or bone marrow after treatment.
Percentage of Participants with Dose Modifications | Up to Month 36
  Dose modifications include interruptions during ramp-up and maintenance phase.
Percentage of Participants with Adverse Drug Reactions (ADR) | Up to Month 36
  ADR is defined as a response to a medicinal product that is noxious and unintended and that a causal relationship between a medicinal product and an adverse event is possible, probable or very likely as assessed by the investigator.
Number of Lines of Prior Therapy in Participants with Relapse/Refractory Chronic Lymphocytic Leukemia | Up to Month 36
  Number of lines of prior therapy per participant, in participants with Relapse/Refractory Chronic Lymphocytic Leukemia.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (21):
- Greece (21):
  - Henry Dunnant Hospital Center /ID# 241682, Athens, Attica
  - General Hospital of Athens Gennimatas /ID# 212917, Athens, Attica
  - General Hospital of Athens Laiko /ID# 212902, Athens, Attica
  - General Hospital of Athens Laiko /ID# 230222, Athens, Attica
  - University General Hospital Attikon /ID# 212915, Athens, Attica
  - Metropolitan General /ID# 212934, Cholargós, Attica
  - Iatriko Kentro Athinon /ID# 241689, Marousi, Attica
  - Iatriko Kentro Athinon /ID# 241690, Marousi, Attica
  - Metropolitan Hospital /ID# 241687, Piraeus, Attica
  - General Hospital of Chania "Agios Georgios" /ID# 241685, Chania, Chania
  - University General Hospital of Heraklion PA.G.N.I /ID# 212916, Heraklion, Crete
  - University General Hospital of Ioannina /ID# 212936, Ioannina, Ioannina
  - Reg Gen Univ Hosp Larissa /ID# 213708, Larissa, Larisa
  - Theageneio Anticancer Hospital /ID# 212933, Thessaloniki, Thessaloniki
  - General Hospital of Thessaloniki George Papanikolaou /ID# 213709, Thessaloniki, Thessaloniki
  - General University Hospital of Alexandroupolis /ID# 212927, Alexandroupoli
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 212929, Athens
  - General Hospital of Patras Agios Andreas /ID# 213711, Pátrai
  - University Gen Hosp of Patra /ID# 212914, Pátrai
  - METAXA Cancer Hospital of Piraeus /ID# 212918, Piraeus
  - Papageorgiou General Hospital /ID# 213710, Thessaloniki

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.rxabbvie.com/